CLINICAL TRIAL: NCT01518803
Title: Influence of a Mediterranean-style Breakfast on Postprandial Lipid Disorders and Inflammatory Processes in Obese Pre-adolescents and Adults
Brief Title: A Mediterranean-style Breakfast and Postprandial Lipid Disorders in Obese Pre-adolescents and Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Javier Sánchez Perona, Tenured Scientist, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AGL2011-23810
Record Dates: First submitted 2012-01-23; First posted 2012-01-26 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Obesity
Keywords: Obesity; Adolescence; Lipid metabolism; Mediterranean diet; Chylomicron; Macrophages
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mediterranean-style breakfast (Active Comparator)
  Interventions: Dietary Supplement: Mediterranean-style breakfast
- Western-style breakfast (Active Comparator)
  Interventions: Dietary Supplement: Western-style breakfast

INTERVENTIONS:
Dietary Supplement: Mediterranean-style breakfast — The experimental meal will be administered early in the morning as breakfast, "Cardioliva" olive oil, bread (2 slices), tomatoes (half piece), fruit juice (200 mL), skim milk (150 mL). The amount of fat administered will be the equivalent to 0.75 g per kg of body weight.
  Arms: Mediterranean-style breakfast
Dietary Supplement: Western-style breakfast — The experimental meal will be administered early in the morning as breakfast, containing butter, bread 82 slices), chocolate milk (200 mL). The amount of fat administered will be the equivalent to 0.75 g per kg of body weight.
  Arms: Western-style breakfast

SUMMARY:
Obesity has a major impact on the development of cardiovascular disease and other related conditions and it is of particular concern in children. The prevalence of childhood overweight and obesity in Spain is among the highest in the European continent. Childhood obesity has been associated with diseases that were thought to apply only to adults, such as the metabolic syndrome. Insulin resistance is the most important risk factor in subjects with severe obesity, which together with visceral obesity, exacerbates postprandial triglyceridemia, increasing cardiovascular risk.

In this context, the investigators hypothesize that the postprandial lipid metabolism is also impaired in obese pre-adolescents, as it is in obese adults. This includes not only exacerbated postprandial triglyceridemia, but also impaired levels of inflammation markers. In addition, the investigators hypothesize that the lipid and protein composition of postprandial chylomicrons and chylomicron remnants are also altered in obese children when compared with their normal-weight counterparts, and that these postprandial lipoproteins induce foam cell formation differently. The investigators also believe that a Mediterranean-style meal can help to normalize the altered postprandial lipid metabolism in obese adolescents.

DETAILED DESCRIPTION:
Excess of body weight has led the World Health Organization to call it a global epidemic. Obesity has a major impact on the development of cardiovascular disease and other related conditions and it is of particular concern in children.

The prevalence of childhood overweight and obesity in Spain is among the highest in the European continent. The health consequences of obesity in children are not as evident as in adults, but childhood obesity has been associated with diseases that were thought to apply only to adults, such as the metabolic syndrome. Insulin resistance is the most important risk factor in subjects with severe obesity, which together with visceral obesity, exacerbates postprandial triglyceridemia, increasing cardiovascular risk.

However, this has not been appropriately studied in children for the moment. The excellent results of previous projects carried out by our research group have shown the beneficial properties of olive oil on health, being the main ingredient of the Mediterranean Diet, including an improved postprandial lipid pattern.

In this context, our hypothesis is that the postprandial lipid metabolism is also impaired in obese pre-adolescents, as it is in obese adults. This includes not only exacerbated postprandial triglyceridemia, but also impaired levels of inflammation markers. In addition, we hypothesize that the lipid and protein composition of postprandial chylomicrons and chylomicron remnants are also altered in obese children when compared with their normal-weight counterparts, and that these postprandial lipoproteins induce foam cell formation differently, as well as a different release of inflammation markers by macrophages. However, it is also part of our hypothesis, that a Mediterranean-style meal,administrated as a breakfast can help to normalize the altered postprandial lipid metabolism in obese children.

With this aim, we will carry out a dietary intervention study with a randomized, crossover design in a single meal, in order to measure changes in the postprandial lipid metabolism in pre-adolescents and adults affected by obesity and to compare the effect of a Mediterranean-style breakfast. Chylomicron remnants will be isolated from blood serum and will be fully characterized. These particles will be incubated with monocyte cell lines to determine their effect on cellular lipid metabolism and the production of inflammatory factors. In addition, the influence of obesity in the composition and structure of the plasma membrane will also be assessed. The results will generate knowledge about the pathophysiology of obesity in children and will contribute to the dietary recommendations for weight maintenance in this population. Furthermore, it will provide information on the development of atherosclerosis during the postprandial period, which may begin at very young ages.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents below 15 years-old with BMI ≥ 30 and above the 95 percentile for their gender and age.
* No history of psychiatric or organic disease, except for obesity.
* Appropriate cultural level to understand the study.
* A written informed consent of their parents or tutors.

Exclusion Criteria:

* Subjects being treated with drugs for any kind of disease.
* Those suffering of chronic diseases.
* A negative to participate in the study from them or their parents or tutors.
* Subjects having participated in another clinical study the preceding 3 months.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2010-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Delay in plasma triglyceride and CM clearance in obese pre-adolescents | 2 and 4 hours postprandially
  It is expected to find a delay in plasma triglyceride and CM clearance in obese pre-adolescents, and to find more atherogenic features in CM and CMR in this group. These characteristics include changes in the lipid and protein composition of lipoproteins. It is expected to define the CM and CMR concentration in the blood of obese pre-adolescents, using as marker the presence of apo B48 in these particles. Particle size and lipid composition will show to what extent CM and CMR are more or less atherogenic in pre-adolescents and obese adults.

SECONDARY OUTCOMES:
Differences in the composition and structure of the plasma membrane in obese volunteers | Time 0, baseline
  We expect to find changes in the composition and structure of the plasma membrane in obese volunteers, which could be related to increased blood pressure. For the first time, we will unravel the molecular species composition of plasma membrane phospholipids of obese pre-adolescents, which will be a milestone in the study of the physiological implications of obesity in this population.

CONTACTS AND LOCATIONS:
Overall Officials: Javier S Perona, PhD, Principal Investigator — National Research Council, Spain
Locations (1):
- Instituto de la Grasa (IG-CSIC), Seville, Seville, Spain

REFERENCES:
- [Background] Aguilar Cordero MJ, Gonzalez Jimenez E, Sanchez Perona J, Padilla Lopez CA, Alvarez Ferre J, Mur Villar N, Rivas Garcia F. [The Guadix study of the effects of a Mediterranean-diet breakfast on the postprandial lipid parameters of overweight and obese pre-adolescents]. Nutr Hosp. 2010 Nov-Dec;25(6):1025-33. Spanish. PMID 21519776